CLINICAL TRIAL: NCT00990067
Title: Pharmacological Interaction Between Duloxetine and 3,4-Methylenedioxymethamphetamine (MDMA, Ecstasy): Pharmacodynamics (PD) and Pharmacokinetics (PK)
Brief Title: Interaction Between Duloxetine and 3,4-Methylenedioxymethamphetamine (MDMA, Ecstasy)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: EKBB 253/09
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Mood Disorder; Substance-Related Disorders; Amphetamine-Related Disorders
Keywords: MDMA; serotonin; norepinephrine; Ecstasy; stimulant
MeSH Terms: conditions — Mood Disorders; Substance-Related Disorders; Amphetamine-Related Disorders | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- duloxetine, MDMA, placebo (Other): Cross-over within-subjects design with all treatment conditions tested in the same subject. This design has 1 arm but two (actually 4) treatment conditions in the same subject.
  Interventions: Drug: 3,4-Methylenedioxymethamphetamine; Drug: Duloxetine; Drug: Placebo

INTERVENTIONS:
Drug: 3,4-Methylenedioxymethamphetamine — 125 mg, single dose
  Other Names: MDMA; Ecstasy
Drug: Duloxetine — 120 mg two doses 12h and 2h before MDMA
  Other Names: Cymbalta (r)
Drug: Placebo — capsules identical to MDMA or duloxetine

SUMMARY:
The purpose of this study is to determinate the effect of a pre-treatment with the combined serotonin (5-HT) and norepinephrine (NE) transport blocker duloxetine on the pharmacodynamics and pharmacokinetics of 3,4-methylenedioxymethamphetamine (MDMA, "Ecstasy"). The investigators hypothesize that duloxetine will attenuate the subjective and cardiovascular response to MDMA.

DETAILED DESCRIPTION:
3,4-methylenedioxymethamphetamine (MDMA, "ecstasy") is widely used by young people for its euphoric effects. MDMA releases serotonin (5-HT), norepinephrine (NE), and dopamine through an interaction with the corresponding presynaptic monoamine uptake transporter. 5-HT transport inhibitors block MDMA-induced 5-HT release in vitro or in animals and also attenuate the subjective and cardiovascular response to MDMA in humans. NE transport inhibitors similarly prevent the MDMA-induced release of NE in cell assays and attenuate behavioral effects of MDMA in animals. Effects of the NE transporter inhibitor reboxetine on the response to MDMA in humans are currently investigated. Here we suggest evaluating effects of pretreatment with the combined 5-HT and NE transport blocker duloxetine on the pharmacodynamics and pharmacokinetics of MDMA. The study will use a randomized double-blind cross-over design with four experimental sessions. Duloxetine (120 mg) or placebo will be administered 16 h and 4 h before the administration of MDMA (125 mg) or placebo to 16 healthy volunteers. Subjective and cardiovascular responses and plasma samples for pharmacokinetics will be repeatedly assessed throughout the experiments.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient understanding of the German language
* Subjects understand the procedures and the risks associated with the study
* Participants must be willing to adhere to the protocol and sign the consent form
* Participants must be willing to refrain from taking illicit psychoactive substances during the study.
* Participants must be willing to drink only alcohol-free liquids and no xanthine-containing liquids (such as coffee, black or green tea, red bull, chocolate) after midnight of the evening before the study session. Subjects must agree not to smoke tobacco for 1 h before and 4 hours after MDMA administration.
* Participants must be willing not to drive a traffic vehicle in the evening of the study day.
* Women of childbearing potential must have a negative pregnancy test at the beginning of the study and must agree to use an effective form of birth control. Pregnancy tests are repeated before each study session.
* Body mass index: 18-25 kg/m2

Exclusion Criteria:

* Chronic or acute medical condition including clinically relevant abnormality in physical exam, laboratory values, or ECG. In particular: Hypertension (>140/90 mmHg). Personal or first-grade history of seizures. Cardiac or neurological disorder.
* Current or previous psychotic or affective disorder
* Psychotic or affective disorder in first-degree relatives
* Prior illicit drug use (except THC (Tetrahydrocannabinol)-containing products) more than 5 times or any time within the previous 2 months.
* Pregnant or nursing women.
* Participation in another clinical trial (currently or within the last 30 days)
* Use of medications that are contraindicated or otherwise interfere with the effects of the study medications (monoamine oxidase inhibitors, antidepressants, sedatives etc.)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Effect of duloxetine on the subjective response to MDMA | 24h

SECONDARY OUTCOMES:
Effect of duloxetine on cardiovascular effects of MDMA | 6h
Effect of duloxetine on pharmacokinetics of MDMA | 6h
Effect of MDMA on duloxetine pharmacokinetics | 6h
Tolerability of MDMA and duloxetine | 7 days
Effect of duloxetine on neuroendocrine responses to MDMA | 6h

OTHER OUTCOMES:
Genetic polymorphisms | assessed after study completion
  Effects of genetic polymorphisms on the response to MDMA

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, Principal Investigator — Department of Internal Medicine, Division of Pharmacology & Toxicology, University Hospital Basel, Switzerland
Locations (1):
- Clinical Pharmacology & Toxicology, University Hospital Basel, Basel, Basel, Switzerland

REFERENCES:
- [Derived] Vizeli P, Liechti ME. Oxytocin receptor gene variations and socio-emotional effects of MDMA: A pooled analysis of controlled studies in healthy subjects. PLoS One. 2018 Jun 18;13(6):e0199384. doi: 10.1371/journal.pone.0199384. eCollection 2018. PMID 29912955
- [Derived] Hysek CM, Liechti ME. Effects of MDMA alone and after pretreatment with reboxetine, duloxetine, clonidine, carvedilol, and doxazosin on pupillary light reflex. Psychopharmacology (Berl). 2012 Dec;224(3):363-76. doi: 10.1007/s00213-012-2761-6. Epub 2012 Jun 15. PMID 22700038
- [Derived] Hysek CM, Simmler LD, Nicola VG, Vischer N, Donzelli M, Krahenbuhl S, Grouzmann E, Huwyler J, Hoener MC, Liechti ME. Duloxetine inhibits effects of MDMA ("ecstasy") in vitro and in humans in a randomized placebo-controlled laboratory study. PLoS One. 2012;7(5):e36476. doi: 10.1371/journal.pone.0036476. Epub 2012 May 4. PMID 22574166
- [Derived] Simmler LD, Hysek CM, Liechti ME. Sex differences in the effects of MDMA (ecstasy) on plasma copeptin in healthy subjects. J Clin Endocrinol Metab. 2011 Sep;96(9):2844-50. doi: 10.1210/jc.2011-1143. Epub 2011 Jun 29. PMID 21715530